CLINICAL TRIAL: NCT06884735
Title: Virtual Reality Exposure Therapy (VRET) for Balance in Patients Suffering from Psychomotor Disadaptation Syndrome
Brief Title: Virtual Reality Exposure Therapy (VRET) in Psychomotor Disadaptation Syndrome
Acronym: TERV-SDPM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-03-TERV-SDPM
Record Dates: First submitted 2025-02-25; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Psychomotor Disadaptation Syndrome
Keywords: Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exposure to a previous vacuum (Experimental): exposure to a previous vacuum
  Interventions: Other: exposure to virtual reality
- museum exposure (Sham Comparator): museum exposure
  Interventions: Other: exposure to virtual reality

INTERVENTIONS:
Other: exposure to virtual reality — exposure to virtual reality

SUMMARY:
According to demographic projections, by 2040, a quarter of the French population will be over 65. In this age group, the quality and quantity of visual, somaesthetic and vestibular information decline. This weakening of the balancing and the recurrence of falls lead to a restriction of activities of daily living and give rise to a fear of falling.

Psychomotor maladjustment syndrome (PMDS) is a serious consequence of falls. A significant retropulsion when sitting or standing, as well as hypertonia characterize the posturobehavioral component of PMDS. It coexists with a psychological component, marked by a fear of the anterior emptiness. A series of studies inducing fear and experimentally manipulating its intensity demonstrated a greater displacement of the center of pressure when subjects were exposed to elevated platforms. In addition to the subjective evaluation of fear, this emotion can be assessed by heart rate variability.

Despite the existence of standards and metrics adapted to the clinical setting, only one study investigated the association between the number of falls and heart rate variability in patients with neurodegenerative disorders. In recent years, cognitive and behavioral therapies using virtual reality (TERV) have improved balance in patients with cardiovascular disease and Parkinson's disease. Virtual reality (VR) thus appears to be an interesting therapeutic approach to the treatment of psychological as well as postural-behavioral disorders of PDMS. Although the feasibility of a VR intervention has been tested in elderly people (APs) suffering from PMDS, its effect has never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PMDS
* Ability to stand without human or technical assistance
* Falls Efficacy Scale International Short (FES-I short) > 13
* Functional Reach Test (FRT) score < 26 cm
* Mini-Mental State Examination (MMSE) score ≥ 20

Exclusion Criteria:

* Patients with disorders that may interfere with immersion in virtual reality (e.g. cerebellar syndromes, Parkinsonian syndromes, hallucinations, sensory or neurocognitive disorders)
* Cybermalaise or cyberkinetosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-03 (Estimated); Study Completion 2028-09-03 (Estimated)

PRIMARY OUTCOMES:
Balance | Day 1
  Average velocity variance of the center of pressure (cm/s) measured by a stabilometric measurement platform before, immediately after, then post-24h exposure to VR

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No